CLINICAL TRIAL: NCT03835819
Title: A Phase 2, Two-stage, Study of Mirvetuximab Soravtansine (IMGN853) in Combination With Pembrolizumab in Patients With Microsatellite Stable (MSS) Recurrent or Persistent Endometrial Cancer (EC)
Brief Title: A Phase 2 Study of Mirvetuximab Soravtansine (IMGN853) and Pembrolizumab in Endometrial Cancer (EC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: ImmunoGen, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-602
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMGN853 + Pembrolizumab (Experimental): * Pembrolizumab is administered intravenously once every 3 weeks
  * IMGN853 is administered intravenously once every 3 weeks
  Interventions: Drug: Pembrolizumab; Drug: IMGN853

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is an immunotherapy that activates a patient's own immune system to recognize and kill tumor cells
  Other Names: Keytruda
Drug: IMGN853 — Mirvetuximab soravtansine is an antibody-drug conjugate.
  Other Names: Mirvetuximab soravtansine; Elahere

SUMMARY:
This research study is studying a drug combination as a possible treatment for endometrial cancer.

The drugs involved in this study are:

* mirvetuximab soravtansine (IMGN853)
* pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved mirvetuximab soravtansine for this specific disease but it has been approved for other uses.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for this specific disease but it has been approved for other uses.

In this research study, the investigators are studying the combination of mirvetuximab soravtansine and pembrolizumab. Pembrolizumab is an immunotherapy that activates a patient's own immune system to recognize and kill tumor cells. Pembrolizumab by itself may not be enough to kill cancer cells in all people with cancer. In this study, all patients will receive mirvetuximab soravtansine and pembrolizumab. Mirvetuximab soravtansine is an antibody-drug conjugate. That is a type of agent that attaches a chemotherapy drug to a molecule that binds a protein on the outside of cancer cells. The protein targeted by mirvetuximab soravtansine is called folate receptor-alpha (FRα). FRα is expressed on the surface of certain cancers, including endometrial cancer cells. Mirvetuximab soravtansine is expected to kill cancer cells by delivering chemotherapy to cells that have high levels of FRα. To participate in this study, a sample of your tumor was previously tested, and was found to have high levels of FRα. Mirvetuximab soravtansine also may also active immune cells and improve the response to immunotherapies like pembrolizumab.

In this study, the investigators expect to learn whether the combination of pembrolizumab and mirvetuximab soravtansine can shrink endometrial cancers or prevent their growth for at least 6 months. The investigators will also learn more about the side effects patients experience who receive this treatment. The investigators also plan to learn more about which patients are likely to benefit from this treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants must have advanced or recurrent serous endometrial cancer. Patients with mixed histologies/tumors are eligible if the serous component is the dominant histological subtype. In addition, the tumors must be:
* microsatellite stable (MSS) as documented by either intact immunohistochemical (IHC) nuclear expression of the mismatch repair genes MSH2, MSH6, MLH1 and PMS2; or microsatelitte stable by polymerase chain reaction (PCR), next generation sequencing, or other CLIA-approved method;

AND

* FRα positive by central immunohistochemistry (IHC, Section 9.1). If archival tissue does not meet FRα criteria, a fresh biopsy tumor sample may be submitted and used to meet this criterium. If a fresh tumor biopsy cannot be done safely the patient will not be allowed to enroll on this study.

  * Participants must have measurable disease as defined by RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
  * Prior therapy: Patients must have had one, but no more than three lines of chemotherapy for endometrial carcinoma.
* Prior hormonal therapy is allowed (no washout period is required after hormonal therapy) and does not count as a prior line of therapy. Hormonal therapy in combination with CDK4/6 inhibitors or mTOR or other PI3K-pathway inhibitors is allowed and does not count as a line of prior therapy.
* Prior IO therapy targeted to the PD-1/PD-L1 pathway is allowed in up to 19 patients of the total cohort.
* Patients must NOT have received prior therapy with any folate receptor ortholog agents.

  * Age 18 or greater years. Because insufficient dosing or adverse event data are currently available on the use of mirvetuximab soravtansine and pembrolizumab in participants <18 years of age, children are excluded. Endometrial cancer is rare in the pediatric population.
  * ECOG performance status 0 or 1
  * Participants must have normal organ and marrow function as defined below:
* leukocytes ≥3,000/mcL
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin ≥ 9.0 g/dL
* total bilirubin ≤ 1.5 x institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
* creatinine ≤ institutional upper limit of normal OR
* creatinine clearance ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.

  -Time from prior therapy:
* Systemic anti-neoplastic therapy: 5 half-lives or 4 weeks, whichever is shorter. Hormonal therapy is not considered anti-neoplastic therapy.
* Radiotherapy: wide-field radiotherapy (e.g. > 30% of marrow-bearing bones) completed at least 4 weeks, or focal radiation completed at least 2 weeks, prior to starting study treatment

  * The effects of agents used in this study on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during study treatment, and for at least twelve weeks after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
  * Women of child-bearing potential must have a negative serum pregnancy test within 3 days prior to the first dose of study treatment.
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy within 5 half-lives or 4 weeks (whichever is shorter) or radiotherapy within 2 weeks prior to entering the study. Patients completing wide-field radiotherapy (e.g. >30% of marrow-bearing bones) must not have had treatment within 4 weeks prior to entering study. Participants must have recovered from all AEs due to previous therapy to Grade 1 ≤ or baseline, except alopecia. Participants with endocrine-related AEs who are adequately treated with hormone replacement are eligible.
* Participants who are receiving any other investigational agents.
* Participants with prior exposure to IO agents targeting the PD-1/PD-L1 pathway who discontinued therapy due to treatment-related toxicity deemed to be specifically related to IO therapy.
* Required use of folate-containing supplements (e.g. folate deficiency).
* Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to monoclonal antibodies (including antibody drug-conjugates or checkpoint inhibitors).
* Uncontrolled intercurrent illness including, but not limited to, any of the following within 6 months of first study treatment: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled hypertension (≥ Grade 3), hypertensive crisis or hypertensive encephalopathy, uncontrolled cardiac arrhythmias, thrombotic or ischemic stroke, clinically-significant vascular disease (e.g. aortic aneurysm, or dissecting aneurysm), severe aortic stenosis, clinically significant peripheral vascular disease, or ≥ Grade 3 cardiac toxicity following prior chemotherapy, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active or chronic corneal disorder, including but not limited to the following: Sjogren's syndrome, Fuchs corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, and also active ocular conditions requiring on-going treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and acquired monocular vision.
* Serious clinically-relevant active infection, including known HIV infection, varicella-zoster virus, cytomegalovirus infection, has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) or any other known concurrent infectious disease requiring IV antibiotics with within 2 weeks of study enrollment are ineligible because of the potential for immune side effects.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Current or prior use of immunosuppressive medication within 7 days prior to enrollment with the following exceptions to this exclusion criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo-or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Pregnant or nursing women are excluded from this study because effects of agents used in this study on infants or the developing human fetus are unknown
* Presence of other malignancies unless they are considered cured by patient's oncologist

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2027-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Porter, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Northwell Cancer Institute, Lake Success, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 18 participants enrolled, all 18 participants are considered evaluable for assessment. Enrollment was closed before the total accrual goal of 35 was met.
Groups:
- IMGN853 + Pembrolizumab: * Pembrolizumab is administered intravenously once every 3 weeks
  * IMGN853 is administered intravenously once every 3 weeks
  Pembrolizumab: Pembrolizumab is an immunotherapy that activates a patient's own immune system to recognize and kill tumor cells
  IMGN853: Mirvetuximab soravtansine is an antibody-drug conjugate.
Period: Overall Study
Arm/Group | IMGN853 + Pembrolizumab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (5.05)
Age, Continuous [Median (Full Range); unit: years] | 67.2 [62.7 to 78.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Stage at Initial Diagnosis [Count of Participants; unit: Participants] — Staging was based on the FIGO (International Federation of Gynecology and Obstetrics) system. Stage I cancers usually have not grown deeply into nearby tissues. Stage II and III cancers have grown more deeply into nearby tissue and may have spread to lymph nodes. Stage IV cancers have spread to other organs or parts of the body. Higher stages are typically associated with worse outcomes.
  Participants
    Stage I | 5
    Stage II | 0
    Stage III | 7
    Stage IV | 6
ECOG Performance Status [Count of Participants; unit: Participants]
  00 - Fully active | 12
  01 - Restricted | 6
Prior Lines [Count of Participants; unit: Participants]
  1 | 2
  2 | 7
  3 | 5
  4 | 4
Prior Anti-PD-1/PD-L1 Exposure [Count of Participants; unit: Participants]
  IO-exposed (avelumab) | 1
  IO-exposed (dostarlimab) | 1
  IO-exposed (pembrolizumab) | 6
  IO-naïve | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate was determined by the frequency of patients who had objective tumor response, determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI, where objective response represents either a confirmed complete response (CR; disappearance of all target lesions) or a confirmed partial response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters); objective response = CR + PR. The ORR is therefore reported as the percentage of participants who achieved a CR or PR per RECIST v1.1.
Time Frame: 6 months
Population: Among 18 patients, 5 had a confirmed response. Confirmed ORR is 28%, with 95% confidence interval of [ 10%, 53%].
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
percentage of participants | 28 [10 to 53]

2. Primary Outcome: Progression-Free Survival at 6 Months (PFS6)
Description: Progression-free survival at 6 months was determined by the frequency of patients who survived progression-free for at least 6 months after initiating study treatment by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), where disease progression represents at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: 6 months
Population: 4 patients were alive and progression-free at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
Participants | 4

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), where disease progression represents at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The distribution of progression-free times will be estimated using Kaplan-Meier analysis.
Time Frame: Interval from start of treatment to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
months | 2.73 [1.2 to 4.5]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive. The distribution of overall survival times will be estimated using Kaplan-Meier analysis.
Time Frame: Participants are followed for survival status from registration through up to 3 years after removal from study intervention
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
months | 11.3 [3.32 to NA] — Upper bound not reached using the KM method.

5. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) is defined as time from best overall response to the time of disease progression.
Time Frame: Interval from best overall response to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first.
Population: Due to the small number of responses, reporting the confidence interval or interquartile range is not meaningful. Out of the 5 confirmed responders, 2 experienced events (progression or death), while 3 were censored.
Measure: Median (Full Range); unit: months
Arm/Group | IMGN853 + Pembrolizumab
Number analyzed (Participants) | 18
months | 7.1 [2.76 to 18.14]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for all participants through 30 days after last intervention (up to 21 months).
Arm/Group | IMGN853 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 12/18
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMGN853 + Pembrolizumab (N=18)
Corneal ulcer (Eye disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Malignant neoplasm of the skin - squamous cell carcinoma
Platelet count decreased (Investigations) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMGN853 + Pembrolizumab (N=18)
Anemia (Blood and lymphatic system disorders) | 10
Sinus tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 8
Cataract (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1 — Corneal microcysts
Photophobia (Eye disorders) | 1
Abdominal distention (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Ascites (Gastrointestinal disorders) | 1
Belching (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Diverticulitis
Hemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 13
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Intermittent shakiness
Generalized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Bacteremia (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Creatinine increased (Investigations) | 6
Fibrinogen decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 8
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Glucose intolerance (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysarthia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 — Vaginal bleeding
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Keratitis (Eye disorders) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 — Arm wound from excision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03835819/Prot_SAP_000.pdf